CLINICAL TRIAL: NCT05806242
Title: EMS-I: Validation of the Italian Version of the Elderly Mobility Scale
Acronym: EMS-I
Status: Completed | Type: Observational
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Responsible Party: Sponsor
Other Study IDs: INRCA_003_2023
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-03

CONDITIONS: Physical Functional Performance
Keywords: elderly subjects; rehabilitation; Elderly Mobility Scale

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Validation: Elderly in-patients eligible for physiotherapy admitted to IRCCS-INRCA Hospital
  Interventions: Other: Italian Validation of the Italian Elderly Mobility Scale (EMS-I)

INTERVENTIONS:
Other: Italian Validation of the Italian Elderly Mobility Scale (EMS-I) — Two physiotherapists independently evaluate the same enrolled patient with the Italian Elderly Mobility Scale (EMS-I) and Barthel Index

SUMMARY:
This study is an observational study that aims to validate the Elderly Mobility Scale (EMS) in Italian (EMS-I) by comparison with the Barthel Index scale, already validated in Italian. Furthermore this study wants to evaluate the inter-rater reliability comparing the scores assigned to the same sample of patients by two independent evaluators. The study population includes 50 elderly in-patients eligible for physiotherapy.

DETAILED DESCRIPTION:
This study is an observational study that aims to validate the Elderly Mobility Scale (EMS) in Italian (EMS-I) by comparison with the Barthel Index scale, already validated in Italian.

The Elderly Mobility Scale (EMS) is considered a suitable tool to assess basic motor function in hospitalized geriatric patients. It has shown good psychometric characteristics.

The study process requires a standardized translation protocol, including forward and backward translation. The protocol provides enrollment of 50 geriatric in-patients eligible for physiotherapy admitted to IRCCS-INRCA Hospital. Two physiotherapists independently evaluate the same enrolled patient with Italian EMS (EMS-I) and Barthel Index.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the IRCCS-INRCA Hospital
* Request for physiotherapy evaluation
* Sign of the informed consent

Exclusion Criteria:

* Lack of Medical approval for sitting and standing position.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Elderly frail in-patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Italian Elderly Mobility Scale (EMS) in Italian (EMS-I) validity | baseline
  Elderly Mobility Scale (EMS) is a validated assessment tool test used by physiotherapists to assess the level of mobility in frail older adults. The total score ranges from 0 (totally dependent) to 20 (independent mobility). The Italian version (EMS-I) has required a standardized translation protocol, including forward and backward translation. EMS-I will be validated by comparison with the Barthel Index scale, already validated in Italian.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS INRCA Hospital, Ancona, Italy

REFERENCES:
- [Derived] Nicolai M, Casoni E, Bertino E, David L, Polverigiani C, Mallucci F, Fioretti P, Leonzi S, Bevilacqua R, Barbarossa F, Maranesi E, Baccini M, Barboni I, Riccardi GR. Evaluation of the Italian version of the elderly mobility scale in older hospitalized patients. Front Public Health. 2023 Nov 15;11:1274047. doi: 10.3389/fpubh.2023.1274047. eCollection 2023. PMID 38035291